CLINICAL TRIAL: NCT06206096
Title: PD-1 Antibody Plus Bevacizumab and CAPOX as First-line Treatment for Patients With RAS-mutant, Microsatellite Stable, Metastatic Colorectal Cancer: a Prospective, Open-label, Single-arm, Phase II Trial
Brief Title: PD-1 Antibody Plus Bevacizumab and CAPOX as First-line Treatment for RAS-mut MSS mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLNK-CRC-01
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; RAS Mutation; Colorectal Neoplasms; Microsatellite Stable Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPOX+BEV+PD-1 (Experimental)
  Interventions: Drug: oxaliplatin+capecitabine+bevacizumab+PD-1 antibody

INTERVENTIONS:
Drug: oxaliplatin+capecitabine+bevacizumab+PD-1 antibody — oxaliplatin will be administered once every 3 weeks at a dose of 130 mg/m2; Capecitabine will be taken orally at a dose of 1g/m2 twice daily for continuous oral administration over 14 days; Bevacizumab will be administered intravenously every 3 weeks at a dose of 7.5 mg/kg; PD-1 antibody was given due to different types.

SUMMARY:
This study is designed to explore the efficacy and safety of anti-PD-1 antibody plus bevacizumab and chemotherapy as first-line treatment for patients with RAS-mutant, microsatellite stable, metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non resectable, locally advanced or metastatic colorectal cancer;
* No previous anti-tumor treatment for metastatic diseases;
* KRAS/NRAS mutation;
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 3 months;
* Adequate organ and bone marrow functions:

Absolute neutrophil count≥1.5x10^9/L; Platelet count≥100x10^9/L; Hemoglobin≥9g/dL; Serum bilirubin<1.5x the upper limit of normal(ULN); Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)<1.5x ULN; Serum creatinine<1.5x ULN; Endogenous creatinine clearance rate ≥ 50ml / min;

* Women of childbearing age need to take effective contraceptive measures.

Exclusion Criteria:

* Previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors or previous use of immune checkpoint inhibitors;
* With BRAF mutation or MSI-H status;
* Other untreated or concurrent tumors (except cervical carcinoma in situ, treated basal cell carcinoma or superficial bladder tumor, or if the tumor is cured and there is no evidence of disease for more than 3 years);
* Have received other systemic anti-tumor treatments, including chemotherapy, signal transduction inhibitors, hormone therapy and immunotherapy within 4 weeks before enrollment;
* There was central nervous system (CNS) metastasis or previous brain metastasis before enrollment;
* Have received any surgery or invasive treatment or operation within 4 weeks before enrollment;
* Have received Local anti-tumor therapy such as hepatic artery interventional embolization, liver metastasis cryoablation or radiofrequency ablation within 4 weeks before enrollment;
* Uncontrolled malignant ascites;
* Participated in other clinical trials within 4 weeks before enrollment, and received corresponding experimental drug treatment;
* Allergic to the study drug or any of its adjuvants;
* International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN；
* The researchers judged clinically significant electrolyte abnormalities;
* Hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg; Patients currently have poorly controlled diabetes (fasting glucose level is greater than CTCAE grade 2 after regular treatment);
* Patients with dysphagia, active peptic ulcer, intestinal obstruction, active gastrointestinal bleeding, peptic perforation, malabsorption syndrome or uncontrolled intestinal inflammatory diseases;
* Any disease or state affecting drug absorption before enrollment, or the patient cannot take oral medication;
* Patients with obvious evidence of bleeding tendency or medical history within 3 months before enrollment, hemoptysis or thromboembolism within 12 months;
* Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%;
* Active infection or serious infection that is not controlled by drug (≥CTCAE v5.0 Grade 2）;
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×10^4/ml or >2000 IU/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×10^3/m); hepatitis and cirrhosis;
* Women who are pregnant or lactating;
* Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0g;
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions that makes the subject not suitable for enrolling according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  The proportion of patients with a confirmed complete response or partial response

SECONDARY OUTCOMES:
PFS | up to 3 years
  The time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first
OS | up to 3 years
  The time from randomization to death from any reason
DCR | up to 3 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD)
Safety and tolerability by incidence, severity and outcome of adverse events | up to 3 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Jia R, Si H, Ma Y, Fan M, Zhang N, Liu F, Shi Y, Jia Y, Zhang Y, Han Q, Wang Z, Dai G. Efficacy and safety of sintilimab plus bevacizumab and CAPOX as first-line treatment for patients with RAS-mutant, microsatellite stable, metastatic colorectal cancer. BMC Cancer. 2025 Mar 7;25(1):422. doi: 10.1186/s12885-025-13794-w. PMID 40055652